CLINICAL TRIAL: NCT03171233
Title: Immediate Effects of Two Ankle Mobilization Techniques in the Amplitude of Dorsiflexion and Dynamic Valgus Knee: a Random Clinical Test
Brief Title: Immediate Effects of Two Ankle Mobilization Techniques in the Amplitude of Dorsiflexion and Dynamic Valgus Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, Master, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCC_Fernanda
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Ankle Joint Contracture; Knee Injuries and Disorders
MeSH Terms: conditions — Knee Injuries; Disease | interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group mobilization with movement (Active Comparator): Techniques to improve ankle mobility that possibily will to cause changes in the biomechanical motion of the lower limb. The patient does the movement actively, but is assisted by the therapist to mobilize.
  Interventions: Other: Mobilization with movement
- Group Self mobilization with movement (Active Comparator): Techniques to improve ankle mobility that possibily will to cause changes in the biomechanical motion of the lower limb. The patient performs the movement and the mobilization in an independently way without receiving help from the therapist
  Interventions: Other: Self mobilization with movement

INTERVENTIONS:
Other: Mobilization with movement — Participants Mobilization Group with Movement are positioned knee facing the physiotherapist, are not elastic passages above the participant's malleolus and are from the physiotherapist's pelvis. The therapist applies a posterolateral slip sustained to a tibia through the belt, leaning backward, while the talus and forefoot are secured with the space between the thumb and the second finger of the hand of both hands. The participant will be instructed to perform a slow dorsiflexion movement for their maximum amplitude.
  Arms: Group mobilization with movement
Other: Self mobilization with movement — In the Auto Mobilization with Movement group, participants will self-mobilize the ankle on top of a box (15 centimeters with a 10 ° incline), a non-elastic band will pass below the malleoli and the back of the band will be placed in the middle of the other Lower limb, thus mobilizing the talus in the posteroinferior direction, the participant should maintain the force in that direction while making the dorsiflexion movement in closed kinetic chain until returning to the initial position again. Using the same group protocol as the therapist will help.
  Arms: Group Self mobilization with movement

SUMMARY:
Dynamic knee valgus is an inadequate biomechanical movement of multifactorial cause that may expose the individual to various injuries. The range of motion of ankle dorsiflexion is one of the possible influencing factors. This study intends to compare the immediate effect of two techniques on ankle mobility and dynamic knee valgus.

DETAILED DESCRIPTION:
This study aims to verify the immediate effects of ankle mobilization on dynamic knee valgus and to compare two techniques of ankle mobility. It will include 102 lower limbs that present deficit of ankle dorsiflexion and dynamic knee valgus in the same lower limb.

Participants will be divided into two groups, one for ankle mobilization with movement aided by the therapist and another for self mobilization of the ankle. The two intervention groups will do the same protocol, same number of sets, repetitions and rest time.There will be randomisation allocation of individuals in the groups and because of the nature of the interventions only the evaluator may be blind.

The Kolmogorov - Smirnov test is used to verify the data distribution normality. The characterization of the participants is performed by means of descriptive statistical analysis. Parametric or non-parametric tests will be used according to the data distribution normality for comparison between groups at baseline. The evaluator blinding will be tested using the chi -square test by comparing the randomization code with the evaluator opinion. The difference between the groups and their respective confidence intervals will be calculated by linear mixed models using interaction term of "time versus group."

ELIGIBILITY:
Inclusion Criteria:

* Physically active individuals (30 minutes of moderate physical activity at least three times a week with at least 6 months of practice); Men or women ranging in age from 18 to 35 years; (With a value equal to or less than 10 cm in the measuring tape and / or 2 cm difference between the limbs) and dynamic knee valgus (center of the patella surpassing the midpoint between the malleoles ) evaluated by Forward Step Down Test (FSDT).

Exclusion Criteria:

* Patients who present any of these conditions will be excluded from the study: chronic ankle instability, previous surgery on the joints of the foot, ankle, knee, hip or ankle joint injury in the last 2 years that caused more than 1 month of withdrawal; Recent muscular or skeletal injuries that do not allow the exercises to be performed; Severe cardiac conditions or other pathological conditions that make physical therapy impossible.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Range of motion of ankle dorsiflexion Range of motion of ankle dorsiflexion | Immediately after intervention
  Closed kinetic chain evaluation to find the greatest distance between the foot and the wall without compensations
Angle of projection in the frontal plane. | Immediately after intervention
  190/5000 Will be measured during the conduct of the Forward Step-Down Test through 2D-captured footage using a digital camera that will be positioned within 2 meters of the step.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel PL Almeida, MsC, Principal Investigator — Universidade Federal do Ceara
Locations (1):
- Federal University of Ceara, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida GP, Carvalho E Silva AP, Franca FJ, Magalhaes MO, Burke TN, Marques AP. Does anterior knee pain severity and function relate to the frontal plane projection angle and trunk and hip strength in women with patellofemoral pain? J Bodyw Mov Ther. 2015 Jul;19(3):558-64. doi: 10.1016/j.jbmt.2015.01.004. Epub 2015 Jan 26. PMID 26118529
- [Background] Amraee D, Alizadeh MH, Minoonejhad H, Razi M, Amraee GH. Predictor factors for lower extremity malalignment and non-contact anterior cruciate ligament injuries in male athletes. Knee Surg Sports Traumatol Arthrosc. 2017 May;25(5):1625-1631. doi: 10.1007/s00167-015-3926-8. Epub 2015 Dec 24. PMID 26704803
- [Background] Barton CJ, Levinger P, Crossley KM, Webster KE, Menz HB. The relationship between rearfoot, tibial and hip kinematics in individuals with patellofemoral pain syndrome. Clin Biomech (Bristol). 2012 Aug;27(7):702-5. doi: 10.1016/j.clinbiomech.2012.02.007. Epub 2012 Mar 20. PMID 22436492
- [Background] Bell DR, Oates DC, Clark MA, Padua DA. Two- and 3-dimensional knee valgus are reduced after an exercise intervention in young adults with demonstrable valgus during squatting. J Athl Train. 2013 Jul-Aug;48(4):442-9. doi: 10.4085/1062-6050-48.3.16. Epub 2013 May 31. PMID 23724771
- [Background] Bennell KL, Talbot RC, Wajswelner H, Techovanich W, Kelly DH, Hall AJ. Intra-rater and inter-rater reliability of a weight-bearing lunge measure of ankle dorsiflexion. Aust J Physiother. 1998;44(3):175-180. doi: 10.1016/s0004-9514(14)60377-9. PMID 11676731
- [Background] Bittencourt NF, Ocarino JM, Mendonca LD, Hewett TE, Fonseca ST. Foot and hip contributions to high frontal plane knee projection angle in athletes: a classification and regression tree approach. J Orthop Sports Phys Ther. 2012 Dec;42(12):996-1004. doi: 10.2519/jospt.2012.4041. Epub 2012 Sep 18. PMID 22990391
- [Background] Collins N, Teys P, Vicenzino B. The initial effects of a Mulligan's mobilization with movement technique on dorsiflexion and pain in subacute ankle sprains. Man Ther. 2004 May;9(2):77-82. doi: 10.1016/S1356-689X(03)00101-2. PMID 15040966
- [Background] Cronstrom A, Creaby MW, Nae J, Ageberg E. Modifiable Factors Associated with Knee Abduction During Weight-Bearing Activities: A Systematic Review and Meta-Analysis. Sports Med. 2016 Nov;46(11):1647-1662. doi: 10.1007/s40279-016-0519-8. PMID 27048463
- [Background] Dill KE, Begalle RL, Frank BS, Zinder SM, Padua DA. Altered knee and ankle kinematics during squatting in those with limited weight-bearing-lunge ankle-dorsiflexion range of motion. J Athl Train. 2014 Nov-Dec;49(6):723-32. doi: 10.4085/1062-6050-49.3.29. PMID 25144599
- [Background] Exelby L. Peripheral mobilisations with movement. Man Ther. 1996 Jun;1(3):118-126. doi: 10.1054/math.1996.0259. PMID 11440498
- [Background] Fong CM, Blackburn JT, Norcross MF, McGrath M, Padua DA. Ankle-dorsiflexion range of motion and landing biomechanics. J Athl Train. 2011 Jan-Feb;46(1):5-10. doi: 10.4085/1062-6050-46.1.5. PMID 21214345
- [Background] Hoch MC, McKeon PO. The effectiveness of mobilization with movement at improving dorsiflexion after ankle sprain. J Sport Rehabil. 2010 May;19(2):226-32. doi: 10.1123/jsr.19.2.226. PMID 20543222
- [Background] Jeon IC, Kwon OY, Yi CH, Cynn HS, Hwang UJ. Ankle-Dorsiflexion Range of Motion After Ankle Self-Stretching Using a Strap. J Athl Train. 2015 Dec;50(12):1226-32. doi: 10.4085/1062-6050-51.1.01. Epub 2015 Dec 3. PMID 26633750
- [Background] Loudon JK, Wiesner D, Goist-Foley HL, Asjes C, Loudon KL. Intrarater Reliability of Functional Performance Tests for Subjects With Patellofemoral Pain Syndrome. J Athl Train. 2002 Sep;37(3):256-261. PMID 12937582
- [Background] Malliaras P, Cook JL, Kent P. Reduced ankle dorsiflexion range may increase the risk of patellar tendon injury among volleyball players. J Sci Med Sport. 2006 Aug;9(4):304-9. doi: 10.1016/j.jsams.2006.03.015. Epub 2006 May 2. PMID 16672192